CLINICAL TRIAL: NCT06011928
Title: Comparison Of Motor Imagery Focused Pelvic Floor Exercises And Relaxation Exercises For Treating Dysmenorrhea: A Randomized Controlled Study
Brief Title: MOPEXE and RE in Treating Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, assistant professor doctor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UskudarU65
Record Dates: First submitted 2023-08-03; First posted 2023-08-25 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Dysmenorrhea; Gynecologic Disease
Keywords: Dysmenorrhea; Menstrual symptom; Imagination; Relaxation; Pelvic floor exercises; exercise
MeSH Terms: conditions — Dysmenorrhea; Genital Diseases, Female; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor imagery focused pelvic floor exercise (MOPEXE) (Active Comparator): Internal imagery technique, one of the imagery techniques, will be applied to the participants.
  Exercise program 8 weeks, 3 days a week, 3 sets of 10 repetitions of each movement and between sets It is planned to rest for 10 seconds.
  Interventions: Other: MOPEX Exercise
- Relaxation exercise (RE) group (Active Comparator): One of the relaxation methods, Progressive Relaxation Exercises will be used.Exercises will be required to be applied 3 days a week, as 1 set of 10 repetitions per day.
  Interventions: Other: Relaxation Exercise
- Combined exercise group (CEG) (Active Comparator): With the video home exercise program, the participants performed progressive relaxation exercises, respectively. then they will be provided with motor imagery focused pelvic floor exercises. A rest period of 5 minutes will be applied between two different exercise programs.
  Interventions: Other: Combine Exercise

INTERVENTIONS:
Other: MOPEX Exercise — Exercises to be done in order:
  1. Pelvic tilt in supine position
  2. Bridge building
  3. Pelvic stretching
  4. Ball spin
  5. Cat-camel exercise
  Exercise program 8 weeks, 3 days a week, 3 sets of 10 repetitions of each movement and between sets It is planned to rest for 10 seconds
  Arms: Motor imagery focused pelvic floor exercise (MOPEXE)
Other: Relaxation Exercise — Progressive muscle relaxation exercises, respectively, facial muscles, neck and shoulders, right-left arm, right-left hand, back muscles, chest muscles, abdominal muscles, hip, right-left leg, right-left foot muscles are contracted while breathing deeply and slowly, and relaxing when exhaling. will be displayed. Each muscle is contracted for 5 seconds and relaxed for 10 seconds. will be held. Before moving on to the new muscle group in intermuscular contraction and relaxation, several times in between Slow and deep breathing will be practiced. After all the muscles are contracted and relaxed in sequence, Then, while inhaling, all the muscles contract simultaneously and while exhaling, will be loosened.
  Arms: Relaxation exercise (RE) group
Other: Combine Exercise — Exercises to be done in order:
  Pelvic tilt in supine position Bridge building Pelvic stretching Ball spin Cat-camel exercise Exercise program 8 weeks, 3 days a week, 3 sets of 10 repetitions of each movement and between sets It is planned to rest for 10 seconds.
  Progressive muscle relaxation exercises, respectively, facial muscles, neck and shoulders, right-left arm, right-left hand, back muscles, chest muscles, abdominal muscles, hip, right-left leg, right-left foot muscles are contracted while breathing deeply and slowly, and relaxing when exhaling. will be displayed. Each muscle is contracted for 5 seconds and relaxed for 10 seconds. will be held. Before moving on to the new muscle group in intermuscular contraction and relaxation, several times in between Slow and deep breathing will be practiced. After all the muscles are contracted and relaxed in sequence, Then, while inhaling, all the muscles contract simultaneously and while exhaling, will be loosened.
  Arms: Combined exercise group (CEG)

SUMMARY:
The aim of this study is to compare the effects of motor imagery focused pelvic floor exercises and relaxation exercises used in the treatment of dysmenorrhea on pain and menstrual symptoms.

DETAILED DESCRIPTION:
Quantitative research methods were used in the study and it was a randomized type study. The sample of the study consisted of women between the ages of 18-30 who volunteered to participate in the study, showed symptoms of dysmenorrhea and can be accessed online. The names of female participants who volunteered to participate in the study and met the inclusion criteria were written on papers and put in a bag. Papers will be randomly selected by the evaluator by drawing lots. Participants will be randomly divided into 3 groups: motor imagery focused pelvic floor exercise group, relaxation exercise group, and combined group. Among the participants who agreed to participate in the study, the sociodemographic and menstrual characteristics information form and the Visual Analogue Scale value of 5 and above on the day when the menstrual cycle is most severe were included in the study, and the McGill Pain Questionnaire-Short Form, Menstruation Attitude Scale (MBI), Functional and Emotional Dysmenorrhea Scale (FEDS) they will be asked to fill in. After the groups are formed, video home exercise programs will be delivered online (whatsApp, mail, etc.) to the participants. Individuals will be asked to apply the created video home exercise program individually in their own environment. Before the participants start their exercise programs, exercise programs will be taught by online interview. You will be asked to do the exercises for 8 weeks, 3 days a week. After the 8-week exercise program is over, the participants will be asked to fill in the McGill Pain Questionnaire- Short Form, Menstruation Attitude Scale (MBI), Functional and Emotional Dysmenorrhea Scale (FEDS) on the day when the menstrual pain is most severe. Pre- and post-intervention data were statistically analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Having a normal menstrual cycle (24-35 days),
* never having given birth
* According to the Visual Analogue Scale (VAS), the pain level during the menstruation period is 10.
* to give a score of 5 or more out of cooperative and oriented
* Volunteer to participate in the study.

Exclusion Criteria:

* Having an active sexual life
* Receiving psychiatric treatment for stress disorder or anxiety, using birth control pills,
* Those with irregular menstrual cycles (less than 21 days or longer than 35 days)
* those with a menstrual cycle period),
* undergoing any gynecological surgery,
* A mental, cardiovascular, pulmonary, or orthopedic disorder that may interfere with exercise have a disease

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — dysmenorrhea is a female disease
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 10 weeks
  The VAS was used on the most severe day of the menstrual cycle to determine the severity of pain, which is one of the inclusion criteria of the participants before starting the study. Subjects were asked to mark the degree of pain they felt on a straight line of 100 millimeters (mm). A 0 at the beginning means no pain and a maximum of 10 at the end of the line means unbearable pain. The point determined on the line expresses the intensity of pain that people feel during menstruation.
McGill pain questionnaire- short form | 10 weeks
  It is a questionnaire used to describe the severity and quality of the pain that a person feels during menstruation. A high score indicates a high level of pain. The questionnaire consists of three parts. In the first part, there are 15 descriptive word groups, 11 of which are to evaluate the emotional/perceptual dimension of pain and 4 to evaluate the emotional/emotional dimension of pain. Words are rated from 0 to 3 (0= None at all, 1= Mild, 2=Moderate, 3= Severe). In the first part, three pain scores are obtained: sensory pain score, perceptual pain score and total pain score. Pain quality scores are obtained with sensory/perceptual 0-33 points, emotional/emotional 0-12 points, and a total of 0-45 points. The second part is the display of the pain intensity of his work on a scale. A low value indicates a low level of pain, and a high value indicates severe. The third section has five word groups ranging from 'mild pain' to 'unbearable pain' to describe one's pain.
Menstruation attitude scale (MBI) | 10 weeks
  It is used to evaluate the positive / negative aspects of menstruation. The scale is a Likert-type scale consisting of 33 items and five subscales. The subscales and the items of the subscales are as follows:
  * Menstruation as a debilitating phenomenon (12 items),
  * Menstruation as a disturbing phenomenon (6 items),
  * Menstruation as a natural phenomenon (5 items),
  * Noticing/anticipating that menstruation will occur (5 items),
  * Denial of the effects of menstruation (7 items) The scale is evaluated by scoring between 1 and 7, and the Turkish form has been converted into scoring between 1 and 5. Participants are asked to mark the most appropriate option (1. Strongly disagree, 2. Disagree, 3. Undecided, 4. Agree, 5. Totally agree).
Functional and emotional dysmenorrhea scale (FEDS) | 10 weeks
  Evaluates dysmenorrhea functionally and emotionally. It consists of 14 items and 2 sub-dimensions. In the scale, each item is scored between 1 and 5 (1. Not at all similar to my situation, 2. Not similar to my situation, 3. Similar or not similar to my situation, 4. Considered similar to my situation, 5. Very similar to my situation). The presence of a high score indicates that the level of functional and emotional impact of dysmenorrhea is high.

CONTACTS AND LOCATIONS:
Overall Officials: Selda KOÇOĞLU, Study Chair — Uskudar University
Locations (1):
- Üsküdar Unıversıty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McKenna KA, Fogleman CD. Dysmenorrhea. Am Fam Physician. 2021 Aug 1;104(2):164-170. PMID 34383437
- [Background] Boztas Elverisli G, Armagan N, Atilgan E. Comparison of the efficacy of pharmacological and nonpharmacological treatments in women with primary dysmenorrhea: randomized controlled parallel-group study. Ginekol Pol. 2023;94(9):687-697. doi: 10.5603/GP.a2022.0009. Epub 2022 Apr 14. PMID 35419791
- [Background] Daley AJ. Exercise and primary dysmenorrhoea : a comprehensive and critical review of the literature. Sports Med. 2008;38(8):659-70. doi: 10.2165/00007256-200838080-00004. PMID 18620466
- [Background] Armour M, Ee CC, Naidoo D, Ayati Z, Chalmers KJ, Steel KA, de Manincor MJ, Delshad E. Exercise for dysmenorrhoea. Cochrane Database Syst Rev. 2019 Sep 20;9(9):CD004142. doi: 10.1002/14651858.CD004142.pub4. PMID 31538328
- [Background] Fuentes-Aparicio L, Cuenca-Martinez F, Munoz-Gomez E, Molla-Casanova S, Aguilar-Rodriguez M, Sempere-Rubio N. Effects of therapeutic exercise in primary dysmenorrhea: an umbrella and mapping review. Pain Med. 2023 Dec 1;24(12):1386-1395. doi: 10.1093/pm/pnad104. PMID 37555833
- [Background] Lopez-Liria R, Torres-Alamo L, Vega-Ramirez FA, Garcia-Luengo AV, Aguilar-Parra JM, Trigueros-Ramos R, Rocamora-Perez P. Efficacy of Physiotherapy Treatment in Primary Dysmenorrhea: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Jul 23;18(15):7832. doi: 10.3390/ijerph18157832. PMID 34360122